CLINICAL TRIAL: NCT01641094
Title: Effect of Telaprevir in Triple Therapy on Intrahepatic Immunological Mechanisms.
Brief Title: Effect of Teleprevir in Triple Therapy on Intrahepatic Immunological Mechanisms
Acronym: ETIM
Status: Completed | Type: Observational
Sponsor: Foundation for Liver Research (Other)
Collaborators: Janssen-Cilag B.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: ETIM
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Hepatitis C
Keywords: Hepatitis C; Liver; Immunology; Genotype 1; Treatment; Chronic; RNA Virus Infections; Ribavirin; Peginterferon alfa-2a; Protease Inhibitors; Telaprevir
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Bronchiolitis Obliterans Syndrome; RNA Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Chronic hepatitis C infection (HCV) is a disease that affects worldwide about 170 million people. The previous standard of care therapy of chronic HCV patients consists of pegylated-IFN-α combined with ribavirin, and results in sustained clearance of HCV-RNA in only about 50% of the HCV genotype 1 infected patients. Telaprevir, a NS3A-4A inhibitor, has previously proven to offer therapeutic options to previous non-responders to the standard of care. Although, not all chronic HCV patients benefit from telaprevir and it is still not known why certain patients are also non-responsive to this triple therapy. In this study we try to understand why certain patients are also non-responsive to telaprevir, how triple therapy modulates the responsiveness to IFN-α and what the immunological consequences are of treatment with telaprevir, either directly or as a result of telaprevir-induced reduction of HCV-RNA levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age, with a chronic hepatitis C - genotype 1 infection
* Patients are naive, non-responders or relapsers to previous treatment with peginterferon or conventional interferon plus ribavirin combination therapy
* High viral load (>400,000 IU/ml)
* Indication for antiviral therapy of hepatitis C according to current clinical guidelines

Exclusion Criteria:

* Decompensated cirrhosis (Child-Pugh Grade B or C)
* Hepatic imaging (ultrasound, CT or MRI) with the evidence of hepatocellular carcinoma.
* Females who are pregnant or breast-feeding
* History or other evidence of severe illness, malignancy or any other condition which would make the patient, in the opinion of the investigators, unsuitable for the study
* Co-infections with human immunodeficiency virus (HIV) or Hepatitis B virus (HBV)
* Presence of contra-indications for antiviral therapy with telaprevir:
* Telaprevir is contraindicated when combined with drugs that are highly dependent on CYP3A for clearance and for which elevated plasma concentrations are associated with serious and/or life-threatening events. Telaprevir in contraindicated when combined with drugs that strongly induce CYP3A and thus may lead to lower exposure and loss of efficacy of Telaprevir. The contraindicated medications include the following:
* Alfuzosin
* Rifampicin
* Dihydroergotamine, ergonovine, ergotamine, methylergonovine
* Cisapride
* St John's wort
* Atorvastatin, lovastatin, simvastatin
* Pimozide
* Sildenafil or tadalafil
* Triazolam
* Presence of contra-indications for antiviral therapy with peginterferon or ribavirin
* Severe psychiatric disorder, such as major psychoses, suicidal ideation, suicidal attempt and/or manifest depression.
* Visual symptoms related to retinal abnormalities
* Pregnancy, breast-feeding or inadequate contraception
* Thalassemia, spherocytosis
* Interfering substance abuse, such as high alcohol intake (indicator: 28 drinks/ week)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C, genotype 1
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Determine functionality of immune cells in the liver and blood in chronic HCV patients before, during and after treatment with telaprevir, pegylated-IFN-a and ribavirin | 24 week follow-up
  By looking at T cells, NK cells and monocytes during triple therapy, as well intrahepatic as in peripheral blood, we try to better understand why some patients respond and others do not respond to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: A. Boonstra, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Netherlands (2):
  - Reinier de Graaf Ziekenhuis, Delft, South Holland
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- See also: Website of the Department of Gastroenterology & Hepatology - Erasmus Medical Center — http://www.gastrolab.nl
- See also: Website of the Erasmus Medical Center Rotterdam — http://www.erasmusmc.nl